CLINICAL TRIAL: NCT03486145
Title: Nitrate-rich Fruit and Vegetable Supplement and Blood Pressure in Normotensive Healthy Young Males: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Nitrate-rich Fruit and Vegetable Supplement on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Karen L. Sweazea (Unknown); Brendan Miller (Unknown)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Director, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AMPED1
Record Dates: First submitted 2017-06-08; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: High Blood Pressure; Flow Mediated Dilation
Keywords: beetroot juice; nitrates and nitrites
MeSH Terms: conditions — Hypertension | interventions — Fruit

STUDY DESIGN:
Intervention Model Description: Participants were stratified by age, height, weight, BMI, blood pressure and athletic status and randomly assigned to consume daily either the fruit and vegetable rich juice supplement (B) or prune juice (A; control treatment).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the study investigators and the participants were blinded regarding supplement assignments, and the identity of the "A" and "B" supplements were not revealed to study investigators until all data analyses were complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FVS (fruit and vegetable juice supplement) (Experimental): The supplement contained ≈ 260-280 mg or 4 mmoles nitrate per two-ounce serving along with ≈ 51 mg total polyphenols. The FVS contains 7880 mg of a proprietary blend of beet root extract (Beta vulgaris), celery stem and leaf extract (Apium graveolens), red spinach leaf extract (Amaranthus dubius), stevia leaf extract (Stevia rebaudiana), and a fruit and vegetable extract blend (green tea leaf, red grape, white grape, bilberry, carrot, grapefruit, papaya, pineapple, strawberry, apple, apricot, cherry, orange, broccoli, green cabbage leaf, onion, garlic, black current, asparagus, tomato, olive and cucumber). Virtually all of the nitrates in FVS derive from the beet, celery, and red spinach extracts.
  Interventions: Dietary Supplement: fruit and vegetable juice supplement
- PRU (prune juice) (Placebo Comparator): The placebo supplement was prune juice (Sunsweet brand 100% prune juice) (PRU). Prune juice was selected based on its very similar caloric and sugar content, its high antioxidant and phenolic profile, but low nitrate content. The prune juice contained <0.6 mg nitrates and 133 mg total polyphenols per two-ounce serving.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fruit and vegetable juice supplement — FVS was provided by Isagenix International LLC in identically sealed bottles labeled labeled "B". Subjects were not told which supplement they received. Each bottle contained one serving (two ounces) of the supplement.
  Arms: FVS (fruit and vegetable juice supplement)
Dietary Supplement: Placebo — PRU was provided by Isagenix International LLC in identically sealed bottles labeled labeled "A". Subjects were not told which supplement they received. Each bottle contained one serving (two ounces) of the supplement.
  Arms: PRU (prune juice)

SUMMARY:
It is hypothesized that the daily supplementation of a nitrate-rich, two-ounce fruit and vegetable energy supplement (Isagenix International LLC) by healthy young adults with a would increase circulating nitrates and improve cardiovascular parameters compared to a nitrate-deficient placebo (prune juice).

DETAILED DESCRIPTION:
Endothelial cells of the peripheral vasculature are key sources of vasoactive factors regulating healthy blood pressure. One of the primary vasodilatory factors released from these cells is nitric oxide (NO). Production of NO is stimulated both through enzymatic-dependent mechanisms via NO synthase, as well as from dietary intake of nitrate-containing foods or supplements that increase NO bioavailability. This study examined whether the daily consumption of a nitrate-rich, two-ounce fruit and vegetable energy supplement (Isagenix International LLC) would increase circulating nitrates and improve cardiovascular parameters compared to a nitrate-deficient placebo (prune juice). Healthy male adults aged 18-40y (n=45) were recruited to participate in this longitudinal double-blind, placebo-controlled, randomized clinical trial. Subjects maintained their typical diet and physical activity patterns during the study. Anthropometric and cardiovascular (blood pressure and flow-mediated dilation (FMD)) parameters, along with plasma nitrates and nitrites were measured at baseline and after one and two weeks of supplementation. Subjects also completed questionnaires on sleep quality and mood. It is hypothesized that the nitrate-rich FVS supplement will provide a good source of dietary nitrates and effectively reduced blood pressure in normotensive, healthy young males.

ELIGIBILITY:
Inclusion Criteria:

• healthy men aged 18-40y

Exclusion Criteria:

* hypo- or hypertension (blood pressure < 100/65 or >140/90
* cigarette use within past year
* food allergies
* specific medication use (nitroglycerin, beta-blockers, calcium channel blockers),
* unwillingness to drink juice concentrates and follow study restrictions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Plasma nitrates and nitrites | Two week change in concentration (week 2 - baseline)
  The primary objective of this study was to examine the short-term effects of a novel, two-ounce nitrate-rich fruit and vegetable supplement (FVS) (AMPED NOx, Isagenix International LLC) on plasma nitrates and nitrites in healthy young men.
Flow-mediated dilation | Two week change in dilation (week 2 - baseline)
  The primary objective of this study was to examine the short-term effects of a novel, two-ounce nitrate-rich fruit and vegetable supplement (FVS) (AMPED NOx, Isagenix International LLC) on endothelial function in healthy young men.
Blood pressure | Two week change in blood pressure (week 2 - baseline)
  The primary objective of this study was to examine the short-term effects of a novel, two-ounce nitrate-rich fruit and vegetable supplement (FVS) (AMPED NOx, Isagenix International LLC) on blood pressure in healthy young men.

SECONDARY OUTCOMES:
Effect of athletic status on endothelial function | Two week change in flow mediated dilation (week 2 - baseline) by athletic status
  To explore whether athletic status modified the flow mediated dilation response to the supplement athletes
Effect of athletic status on blood pressure | Two week change in blood pressure (week 2 - baseline) by athletic status
  To explore whether athletic status modified the blood pressure response to supplementation

OTHER OUTCOMES:
FMD and mood | Two week change in FMD and mood
  The association of FMD with mood
FMD and sleep quality | Two week change in FMD and sleep quality
  The association of FMD with sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sweazea KL, Johnston CS, Miller B, Gumpricht E. Nitrate-Rich Fruit and Vegetable Supplement Reduces Blood Pressure in Normotensive Healthy Young Males without Significantly Altering Flow-Mediated Vasodilation: A Randomized, Double-Blinded, Controlled Trial. J Nutr Metab. 2018 Sep 16;2018:1729653. doi: 10.1155/2018/1729653. eCollection 2018. PMID 30305961